CLINICAL TRIAL: NCT04871295
Title: Randomized, Controlled Trial of a Weight Loss Intervention in Improving Quality of Life in Men and Women With Overweight or Obesity
Brief Title: Improving Quality of Life in Men and Women With Overweight or Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00048812
Record Dates: First submitted 2021-04-06; First posted 2021-05-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Overweight and Obesity; Quality of Life; Health Behavior
MeSH Terms: conditions — Obesity; Overweight; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List (No Intervention)
- Noom Healthy Weight (Experimental)
  Interventions: Behavioral: Noom Healthy Weight

INTERVENTIONS:
Behavioral: Noom Healthy Weight — Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss with 1:1 coaching The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach. Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight and physical activity on a weekly basis, and meals daily.
  Arms: Noom Healthy Weight

SUMMARY:
The purpose of this study is to evaluate the effect of the Noom Healthy Weight Program, a digital behavior change weight loss intervention, on quality of life as measured both by self-report and objective measures, compared to a waitlist control condition.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* 18-65 years old
* Self-report of good health (physical and mental)
* Not diagnosed with diabetes
* Overweight or obesity (BMI ≥ 25)
* Able to meet our criteria of adherence to the program (at least 1 engagement per week on one of the following: logged exercise, logged meals, steps, weigh-ins, coach messages, read articles, and days with at least one weigh-in.)
* For females
* Not within the 6 months postpartum time frame
* Not planning to become pregnant in the next 5 months.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent
* Currently taking medication which affects sleep or heart rate (e.g., (i) central nervous system stimulants, (ii) respiratory medications, (iii) antihistamines, (iv) central acting hormones (e.g. corticosteroids, thyroid), (v) high-dose anticholinergics, (vi) and cannot be using the maximum recommended dose for antihypertensive medications or use of multiple antihypertensive medications)
* Current diagnosed mental health condition (except mild anxious or depressive symptoms)
* Current diagnosed sleep disorder or condition not related to obesity (e.g., narcolepsy)
* Currently pregnant or ≤ 6 months postpartum
* Currently participating in shift work and/or have travelled between time zones in the last month
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the quality of the data; E.g., evidence of an eating disorder, major chronic condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Weight | 4 months
  Self Reported
In app engagement measures | 4 months
  Self reported and automatically recorded
Stress | 4 months
  Measured via heart rate variability; Data will be collected with a wearable tracking device (Oura Ring). Heart rate variability (HRV) measures the specific changes in time (or variability) between successive heart beats. The time between beats is measured in milliseconds (ms) and is called an "R-R interval" or "inter-beat interval (IBI).

SECONDARY OUTCOMES:
Self Reported Perceived Stress | 4 months
  Perceived Stress Scale (PSS) Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Sleep Quality | 4 months
  Pittsburgh Sleep Quality Index (PSQI); The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Sleep Impact | 4 months
  Adult Sickle Cell Quality of Life Measurement (ASCQ-Me); 5 point rating scale ranging from never - always.
Sleep Score | 4 months
  Measured via a wearable health tracking device (Oura Ring). Sleep score consists of: Total sleep time, time in bed, sleep efficiency, and resting heart rate.
Appetite and food craving | 4 months
  Food Cravings Questionnaire-State; he Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items and response categories range from 1 = strongly disagree to 5 = strongly agree
Reward-related eating | 4 months
  Reward based eating scale (RED-9); A validated, 9-item index that captures reward-based eating drive as a single factor
Perceived physical and mental health over time | 4 months
  Reported via the Health-related quality of life (HRQoL) survey; A multi-dimensional concept that includes domains related to physical, mental, emotional, and social functioning. It goes beyond direct measures of population health, life expectancy, and causes of death, and focuses on the impact health status has on quality of life.
  85 = Very good quality of life. 70 = Good quality of life. 57.5 = Moderately good quality of life.
Depression and anxiety | 4 months
  Depression Anxiety Stress Scales (DASS); The DASS is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress.
  Scoring:
  Normal
  Depression: 0-9
  Anxiety: 0-7
  Stress: 0-14
  Mild
  Depression: 10-13
  Anxiety: 8-9
  Stress: 15-18
  Moderate
  Depression: 14-20
  Anxiety: 10-14
  Stress: 19-25
  Severe
  Depression: 21-27
  Anxiety: 15-19
  Stress: 26-33
  Extremely severe
  Depression: 28+
  Anxiety: 20+
  Stress: 34+

OTHER OUTCOMES:
COVID status | 4 months
  COVID health questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No